CLINICAL TRIAL: NCT00041236
Title: Exatecan As Second-Line Treatment In Advanced Adult Soft Tissue Sarcoma: A Phase II - Study Of The EORTC Soft Tissue And Bone Sarcoma Group
Brief Title: Exatecan Mesylate in Treating Patients With Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-62006; EORTC-62006
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Sarcoma
Keywords: adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; stage IV adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult rhabdomyosarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; uterine leiomyosarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Rhabdomyosarcoma | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of exatecan mesylate in treating patients who have advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the anticancer activity of exatecan mesylate, in terms of objective response and duration of response, in patients with advanced soft tissue sarcoma.
* Determine the safety of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to histological diagnosis (leiomyosarcoma vs other histologies).

Patients receive exatecan mesylate IV over 30 minutes daily on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 weeks until disease progression. After disease progression, patients are followed every 12 weeks for survival.

PROJECTED ACCRUAL: A total of 32-50 patients (16-25 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma

  * Malignant fibrous histiocytoma
  * Liposarcoma
  * Rhabdomyosarcoma
  * Synovial sarcoma
  * Malignant paraganglioma
  * Fibrosarcoma
  * Leiomyosarcoma
  * Angiosarcoma including hemangiopericytoma
  * Malignant peripheral nerve sheath tumor
  * Unclassified sarcoma
  * Miscellaneous sarcoma including mixed mesodermal tumors of the uterus
* The following tumor types are excluded:

  * Gastrointestinal stromal tumor
  * Chondrosarcoma
  * Malignant mesothelioma
  * Neuroblastoma
  * Osteosarcoma
  * Ewing's sarcoma
  * Embryonal rhabdomyosarcoma
* Prior chemotherapy for metastatic disease required

  * One line of combination chemotherapy containing anthracycline OR
  * No more than 2 single-agent regimens including anthracycline
  * Adjuvant chemotherapy not considered first line unless tumor progresses within 6 months after treatment
* Must have 1 measurable lesion

  * Clinical evidence of progression within 6 weeks prior to study
  * Osseous lesions and pleural effusions not considered measurable
* No known or symptomatic CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 15 to 75

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.8 mg/dL
* Albumin at least 2.5 g/dL

Renal:

* Creatinine no greater than 1.4 mg/dL OR
* Creatinine clearance greater than 65 mL/min

Cardiovascular:

* No history of severe cardiovascular disease

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 6 months after study participation
* No other severe medical illness, including psychosis
* No other prior or concurrent malignancy except adequately treated basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy
* No other concurrent cytotoxic therapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No radiotherapy to the sole measurable lesion
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No other investigational drugs for 28 days prior to, during, and for 28 days after completion of study drug
* No other concurrent anticancer therapy

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2002-05; Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reichardt, MD, Study Chair — Robert Roessle Klinik
Locations (10):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - U.Z. Gasthuisberg, Leuven
- Aarhus University Hospital - Aarhus Sygehus - Norrebrogade, Aarhus, Denmark
- Germany (6):
  - Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin
  - Universitatsklinikum Carl Gustav Carl Carus, Dresden
  - Universitaetsklinikum Essen, Essen
  - Universitaets-Krankenhaus Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Eberhard Karls Universitaet, Tübingen
- National Cancer Institute - Bratislava, Bratislava, Slovakia

REFERENCES:
- [Result] Reichardt P, Nielsen OS, Bauer S, Hartmann JT, Schoffski P, Christensen TB, Pink D, Daugaard S, Marreaud S, Van Glabbeke M, Blay JY; EORTC Soft Tissue and Bone Sarcoma Group. Exatecan in pretreated adult patients with advanced soft tissue sarcoma: results of a phase II--study of the EORTC Soft Tissue and Bone Sarcoma Group. Eur J Cancer. 2007 Apr;43(6):1017-22. doi: 10.1016/j.ejca.2007.01.014. Epub 2007 Mar 1. PMID 17336054
- [Result] Pink D, Reichardt P, Nielsen OS, et al.: Exatecan (DX-8951f), a new topoisomerase I - inhibitor, is inactive in heavily pretreated patients (pts.) with advanced soft tissue sarcoma (STS): a phase II study of the EORTC Soft Tissue and Bone Sarcoma Group. [Abstract] J Clin Oncol 23 (Suppl 16): A-9058, 830s, 2005.